CLINICAL TRIAL: NCT05568615
Title: Multicenter, Open-label Extension Study Following the Studies MT-1186-A03 or A04 to Evaluate the Safety of Oral Edaravone in Subjects With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Extension Study Following the Studies MT-1186-A03 or A04 to Evaluate the Safety of Oral Edaravone in Subjects With ALS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-1186-A-301; jRCT2041220069 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2022-10-02; First posted 2022-10-05 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: ALS
MeSH Terms: interventions — Edaravone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MT-1186 orally (Experimental): Subjects receive the edaravone oral suspension orally once daily for 10 days out of a 14-day period, followed by a 14-day drug-free period.
  Interventions: Drug: MT-1186

INTERVENTIONS:
Drug: MT-1186 — Suspension
  Other Names: Edaravone

SUMMARY:
The purpose of this study is to evaluate the safety of oral edaravone at a dose of 105 mg administered once daily for 10 days out of a 14-day period, followed by a 14-day drug-free period. This study will be continued until the earlier date when oral edaravone is commercially available at each site in Japan or August 2023.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide a signed and dated informed consent form (ICF) to participate in the study.
* Subjects must be able (in the judgment of the Investigator) to understand the nature of the study and all risks involved with participation in the study
* Subjects must be willing to cooperate and comply with all protocol restrictions and requirements.
* Subjects who successfully complete Week 96 of Study MT-1186-A03 or Week 48 of Study MT-1186-A04 and have been compliant with study drug (80-120%).

Exclusion Criteria:

* Subjects of childbearing potential unwilling to use a highly effective method of contraception from the Visit #1 until 3 months after the last dose of study medication.
* Subjects who have a significant risk of suicide. Subjects with any suicidal behavior or suicidal ideation of type 4 (active suicidal ideation with some intent to act, without a specific plan) or type 5 (active suicidal ideation with specific plan and intent) based on the C-SSRS at Week 96 of the A03 study or at Week 48 of the A04 study.
* Subjects who are not eligible to continue in the study, as judged by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (11):
- Japan (11):
  - National Hospital Organization Higashinagoya National Hospital, Nagoya, Aichi-ken
  - National Hospital Organization Chibahigashi National Hospital, Chiba, Chiba
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - Kitasato University Hospital, Sagamihara-shi, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - National Hospital Organization Kumamoto Saishun Medical Center, Kōshi, Kumamoto
  - National Hospital Organization Osaka Toneyama Medical Center, Toyonaka-shi, Osaka
  - Shiga University of Medical Science Hospital, Ōtsu, Shiga
  - Tokyo Metropolitan Neurological Hospital, Fuchu-shi, Tokyo
  - National Epilepsy Center NHO Shizuoka Institute of Epilepsy and Neurological Disorders, Shizuoka

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- MT-1186: MT-1186 105mg (2weeks On/Off)
Period: Overall Study
Arm/Group | MT-1186
Started | 15
Completed | 13
Not Completed | 2
Not completed — Death | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | MT-1186
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 0
  Black or African American | 0
  Asian - Japanese | 15
  Asian - Not Japanese | 0
  American Indian or Alaska Native | 0
  Native Hawaiian or Other Pacific Islander | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With AEs and Adverse Drug Reactions
Description: Adverse Event (AE) is classified as treatment emergent if it newly occurred after the first dose of investigational product or if a pre-dose event increases in severity following the first dose of investigational product.
  Adverse Drug Reaction (ADR) is a noxious and unintended response to a medicinal product that occurs at doses normally used for prophylaxis, diagnosis, or therapy of disease.
Time Frame: up to 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | MT-1186
Number analyzed (Participants) | 15
Participants
  Number of patients with AEs | 6
  Number of patients with adverse drug reactions | 0

2. Other Pre Specified Outcome: ALSFRS-R Total Score
Description: The ALSFRS-R is rating scale (ratings 0 = can't do, to 4 = normal ability) used to determine participants' assessment of their capability and independence in 12 functional activities.
Time Frame: up to 10 months or 31/Aug/2023
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Number of Death, Tracheostomy, or Permanent Assisted Mechanical Ventilation (≥23 Hours/Day)
Time Frame: up to 10 months or 31/Aug/2023
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 8 months
Description: This study was a single arm open-label study including the following one single set of dosing regimen specified in the study protocol: 28 days per cycle, study drugs were received for 10 days in the first 2 weeks and subsequently were not received for the rest 2 weeks. The dosing regimen was not divided into Treatment Period or Drug-Free Period since this was a single arm study. Therefore, AE were not collected respectively per specific intervention in this study.
Arm/Group | MT-1186
All-Cause Mortality (participants affected / at risk) | 1/15
Serious Adverse Events (participants affected / at risk) | 2/15
Other Adverse Events (participants affected / at risk) | 5/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MT-1186 (N=15)
Pneumonia aspiration (Infections and infestations) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MT-1186 (N=15)
Otitis externa (Infections and infestations) | 1
Tinea cruris (Infections and infestations) | 1
Constipation (Gastrointestinal disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Catheter site granuloma (General disorders) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Vital capacity decreased (Investigations) | 1
Contusion (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/15/NCT05568615/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/15/NCT05568615/SAP_001.pdf